CLINICAL TRIAL: NCT06494384
Title: Type III Hybrid Effectiveness-Implementation Trial of a Clinical Decision Support System for the Implementation of Problem-Solving Treatment in Community Health Centers
Brief Title: Implementation of Problem-Solving Treatment in Community Health Centers (PST-Aid)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Patrick Raue, Professor, Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00020564; P50MH115837-06 (NIH)
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Problem Solving Treatment as usual (PST as usual) (Active Comparator): Participants in this arm will receiving training in PST as usual.
  Interventions: Behavioral: Problem Solving Treatment as usual (PST as usual)
- Problem Solving Treatment Aid (PST-Aid) (Experimental): Participants in this arm will receiving training in PST with PST-Aid.
  Interventions: Behavioral: Problem Solving Treatment Aid (PST-Aid)

INTERVENTIONS:
Behavioral: Problem Solving Treatment as usual (PST as usual) — PST is a skills-based intervention that teaches clients a 7-step approach in which they 1) select a specific problem and define it in concrete terms,2) select a goal that is feasible to reach before next session, 3) brainstorm various ways to accomplish the goal, 4) evaluate pros and cons of each solution, including the likelihood they can actually implement it, 5) select the best solution, 6) create a plan to implement the solution, and 7) evaluate the plan afterward to ascertain the effectiveness of the solution. Practitioners teach and illustrate the PST process to clients at each session and encourage clients to implement action plans developed using the PST process. Clients are also encouraged to practice the PST process with additional problems between sessions, in order to gain mastery over the PST skills, enhance behavioral activation and as a result improve their belief in their ability to solve problems on their own (self efficacy).
  Arms: Problem Solving Treatment as usual (PST as usual)
Behavioral: Problem Solving Treatment Aid (PST-Aid) — PST-Aid is an internet-based tool to support the delivery of PST. PST-Aid incorporates decision support for the practitioner as well as client and provides PST treatment support functions (i.e., scaffolding), including patient problem lists and session worksheets. PST-Aid was designed to be used during remote sessions, such that practitioners and clients can interact throughout the session while collaboratively viewing and editing worksheets on their own browsers.This system was developed into a prototype that was piloted and found to be acceptable and with adequate usability.
  Arms: Problem Solving Treatment Aid (PST-Aid)

SUMMARY:
Although evidence-based clinical interventions (CI) are a preferred treatment option for patients with depression, CIs are rarely available in community primary care settings. When available, CIs are often delivered with poor fidelity and abandoned by practitioners during the initial months post-training. Identifying effective implementation strategies to support the adoption, reach, and sustained use with fidelity of these CIs could enhance the effectiveness of primary care-based treatment of depression, as primary care is where most treatment for this disorder is delivered. Current models of primacy care practitioner training and supervision follow standard formal didactic procedures that might not be sufficient for successful adoption, high-fidelity delivery, and sustainment of CIs. Automated decision support tools and feedback systems embedded in health informatics technology have been found to be effective in supporting the use of best practices and hence might be useful for the transition from training to sustained CI use. In practice, however, these tools are ignored by practitioners, have mixed success on outcomes, and can hinder clinical care owing to poor design. Problem Solving Treatment Aid (PST-Aid), an educate and reorganize implementation strategy, is a web-based app that promotes practitioner-client collaboration in the use of PST for goal setting and action planning. A pilot randomized trial comparing Problem Solving Treatment (PST) training-as-usual to training plus PST-Aid found PST-Aid was deemed to be appropriate and usable to both practitioner and client users with preliminary support for benefits in depression outcomes.

DETAILED DESCRIPTION:
This study is a hybrid type III effectiveness-implementation randomized clinical trial comparing standard PST implementation with PST augmented by the PST-Aid implementation strategy. The study will test whether:

1. PST Aid results in improved implementation outcomes (initial and sustained fidelity, adoption, reach, and reduced reactive adaptations);
2. Changes in usability, engagement, and appropriateness mediate the effect of PST Aid on implementation outcomes; and
3. PST Aid is more effective in reducing client depressive symptoms and improving functioning.

ELIGIBILITY:
Inclusion Criteria:

* Practitioner Participants. (a) are employed by a clinic that is an OCHIN clinical network member;
* Practitioner Participants. (b) hold a master's degree in social work, psychology, counseling, or a related field;
* Practitioner Participants. (c) provide psychotherapeutic care in the OCHIN network;
* Practitioner Participants. (d) have not previously received formal training in PST as defined by University of Washington Advancing Integrated Mental Health Solutions Center (AIMS) criteria;
* Practitioner Participants. (e) are not currently receiving specialized training outside of standard clinic support to implement a depression-specific psychosocial intervention; and
* Practitioner Participants. (f) are English-speaking.
* Client Participants. a) 18+,
* Client Participants. b) English-speaking,
* Client Participants. c) have a diagnosis of unipolar depression per provider report, and
* Client Participants. d) have a PHQ-9 score ≥ 10, which is above the clinical cutoff for depression symptoms.

Exclusion Criteria:

* Client Participants. (a) history or presence of psychiatric diagnoses other than unipolar, nonpsychotic depression or anxiety disorders,
* Client Participants. (b) active suicidal ideation,
* Client Participants. (c) current alcohol or substance abuse disorders, or
* Client Participants. (d) have dementia
* Client Participants. (e) all exclusion criteria cannot be confirmed via provider report.
* Practitioner Participants. Exclusion criteria are those that do not meet the inclusion criteria listed above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Implementation Strategy Usability Scale (ISUS) score | Baseline, 3 months, 6 months
  Usability will be evaluated with clinician report on the 10-item Implementation Strategy Usability Scale (ISUS), which is based closely on the well-validated System Usability Scale. Ratings are on a 1 to 5 scale and yield a total score from 0 to 100. Half the items are reverse scored; higher total scores reflect greater usability. The ISUS has good inter-item consistency (a = .83) and sensitivity. Research has also demonstrated that the original version of the ISUS (the SUS) functions similarly-and yields similar scores-for adults and youth as young as 11 years.
Change in Participant Responsiveness Scale (PRS) score | Baseline, 3 months, 6 months
  Clinicians will complete the Participant Responsiveness Scale (PRS), an adapted version of the 12-item Patient Responsiveness Scale tailored to be developmentally appropriate for children aged 8 and above as well as adults. The PRS measures two factors, Participation and Enthusiasm. The original Patient Responsiveness Scale has demonstrated strong reliability (a = .86) and construct validity.
Change in Intervention Appropriateness Measure (IAM) score | Baseline, 3 months, 6 months
  Clinicians will complete the Intervention Appropriateness Measure (IAM) is a rigorously developed, pragmatic instrument with strong good internal consistency (a = .87) and test-retest reliability (a = .87).
Adoption over time | Baseline, 7 months post-initial training in the intervention, and end of the individual's study participation period, assessed as the study withdrawal date or 24 months post-training, whichever is first
  Adoption is operationalized as whether or not the clinician completes at least 1 PST session with 3 or more cases at any point during study participation.
Reach over time | Baseline, 7 months post-initial training in the intervention, and end of the individual's study participation period, assessed as the study withdrawal date or 24 months post-training, whichever is first
  Reach will be calculated as the percentage of clinicians caseloads of patients with a depressive disorder receiving PST.
Change in Patient Health Questionnaire (PHQ-9) score | Baseline, 4 weeks, 9 weeks
  The Patient Health Questionnaire is one of the most used short depression measures. The PHQ features 9 items on a four-point scale (0=not at all, 1=several days, 2=more than half the days, 3=nearly every day), with cutpoints for 5, 10, 15, and 20 representing mild, moderate, moderately severe, and severe levels of depressive symptoms. Four original validation studies were conducted on nearly 10,000 patients, and there have been multiple meta-analyses. Scores have been found valid, with sensitivity of 88% and specificity of 88% for a cut point of 10 has been found for Major Depressive Disorders.
Client Satisfaction Questionnaire-16 | 9 weeks
  This measure will ask 3 items from the Client Satisfaction Questionnaire-16: Did treatment meet your needs? Are you satisfied with treatment services? Would you use the same treatment again if needed?
Change in Quality of Life in Neurological Disorders Social Relations scale (Neuro-QOL) score | Baseline, 4 weeks, 9 weeks
  The Quality of Life in Neurological Disorders Satisfaction with Social Roles scale (Neuro-QOL) is a widely used 8-item measure of functioning in usual social roles, activities, and responsibilities. Factor analyses and Item Response Theory analyses have ensured broad information parameters without differential item functioning by demographics. Scale scores have been validated and normed on thousands of participants in the US general and clinical inpatient and outpatient settings, presenting with a variety of problem areas. Scores provide a T score with a mean of 50 and standard deviation of 10, aligned with a variety of norming samples. An example item stem is: In the past 7 days I am able to do all of my regular family activities. Response options are on a scale of 1 to 5 (1=never, 2-rarely, 3=sometimes, 4=often, 5=always).
Initial fidelity (PST Fidelity Scale) | Expert clinicians review audiotapes of therapy sessions or mock interview for each clinician participant over a six-month period of time prior to certification in the intervention
  Fidelity will be measured using the PST Adherence and Competency Scale (PST Fidelity Scale). The PST Fidelity Scale includes seven items assessing the seven key problem-solving steps rated on a 5 point scale (0=very poor, 5=very good), an average score of 3 or greater indicates a satisfactory performance.Internal consistency is good, with Cronbach alpha ranging from .83 to .89. A Principal Components Analysis found all factors loaded on a common factor accounting for 76.6% of the variance.Interrater reliability has been found to be high (r=.822-.918), with 86% of two-rater comparisons within one point of each other. Initial fidelity will be defined as the hours of training until fidelity-based certification is reached, measured by trainer PST Fidelity Scale ratings of session recordings or mock interviews.
Sustained fidelity | Expert clinicians review audiotapes of therapy sessions or mock interview for each clinician participant over a six-month period of time after initial training
  Sustained fidelity will be rated via observer coding of recordings of one randomly selected session (or mock interview) per client using the PST Fidelity Scale (i.e., fidelity tool)

SECONDARY OUTCOMES:
Framework for Modifications and Adaptations of Evidence-based Interventions | End of the individual's study participation period, assessed as the study withdrawal date or 24 months post-training, whichever is first
  This measure will document reactive adaptations to the use of the PST-Aid implementation strategy and the unadapted PST implementation strategy. Based on randomization, clinicians will be provided the set of implementation strategies (e.g., Aid vs. the unadapted PST implementation strategy), and this measure will document what they will be able to do with the goal of understanding some of the natural refinements and adaptations to the implementation strategy. The Framework for Modifications and Adaptations of Evidence-based interventions (FRAME), the leading method for evaluating the nature of intervention adaptations will be used.
Quality of goal setting and action planning over time | Baseline, 4 weeks, 9 weeks
  Using observations of audio recorded sessions, coders will complete the PST Adherence Scale, a seven-item measure scored on a 0 to 5 scale (0=very poor, 5=very good). Six items assess fidelity to technical skills and completing the six specific problem-solving stages. Cronbach alpha coefficients range from .83 to .89. Average item-level interrater agreement is 86%. A seventh item provides a global rating of overall clinician performance, accounting for patient and problem complexity.
Costs over time | Baseline, 3 months, 6 months, 12 months
  A cost checklist will be built for (1) trainers, (2) trainees, and (3) clinics. Participants will estimate the amount of time they spend on conducting PST-related training, meetings, treatment, and providing materials and other costs.
Change in PST Task Self Efficacy Scale score | Baseline, 4 weeks, 9 weeks
  Clients will complete the PST Task Self Efficacy scale, which is based on guidelines for task-specific reliable and valid measures of Task Self Efficacy. Items are on a scale from 0-100 with the stem: Rate your degree of confidence in your ability to do the following. Items are keyed to the specific actions in PST such as defining a problem in their lives connected to depression, establishing realistic goals, and generating solutions. This approach to generating action-specific (task) self-efficacy measures has been successfully used by hundreds of research projects, and is theoretically more internally valid for a study than standardized general measures of self-efficacy.
Change in Behavioral Activation for Depression Scale score | Baseline, 4 weeks, 9 weeks
  Clients will complete the Behavioral Activation for Depression Scale, a 25-item measure on a scale from 0 (not at all) to 6 (completely), which tracks changes in behaviors that underlie depression in the following areas: activation, avoidance/rumination, work/school impairment, and social impairment.Total score and subscale internal consistencies range from .78 to .87. Construct validity has been established with correlations in expected directions with the Beck Depression Inventory, Beck Anxiety Inventory, and Interpersonal Events Schedule.
Change in General Anxiety Disorder-7 (GAD-7) score | Baseline, 4 weeks, 9 weeks
  The General Anxiety Disorder-7 is a seven-item measure on a four-point scale (0=not at all, 1=several days, 2=more than half the days,3=nearly every day), with cutpoints for 5, 10, and15 representing mild, moderate, and severe levels of anxiety symptoms. Scores have been found valid, at the cutpoint of 10 sensitivity and specificity exceeds .80 for Generalized Anxiety Disorder diagnoses. Concurrent validity has been found with positive associations with the Beck Anxiety Inventory and other anxiety scales. Factor analyses have confirmed anxiety items from the GAD as a separate dimension from depression items on the PHQ.
Top Problems Assessment over time | Baseline, 4 weeks, 9 weeks
  The Top Problems Assessment (TPA) is an assessment in which clients are asked to list the problems they are most concerned about. Upon completion of the list, respondents are asked to assign a severity rating for each problem by answering the questions: how big of a problem is this for you? (0 = not at all to 10 =very, very much). Respondents are then asked to identify which of the problems listed is the biggest problem right now? Which one is the most important to work on? Then the second and third most important until 3 top problems are identified.The TPA is an unchanged version of the Youth Top Problems Assessment (YTPA), which shows excellent concurrence with standardized assessments (Kappa ranging from .78 to .91), while also adding specificity for treatment targets. While the TPA has not yet been validated using an adult sample, the wording is applicable to all age ranges and there is all rationale supports the appropriateness of its usage.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Raue, PhD, Principal Investigator — University of Washington
Locations (1):
- OCHIN, Inc., Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No